CLINICAL TRIAL: NCT03966339
Title: Growth Hormone Adding to Controlled Ovarian Hyperstimulation for Improving Embryo Quality：a Randomized Controlled Study
Brief Title: Growth Hormone Adding to Controlled Ovarian Hyperstimulation for Improving Embryo Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2019004
Record Dates: First submitted 2019-05-14; First posted 2019-05-29 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Infertility,Female
Keywords: Infertility,Female; Embryo Development
MeSH Terms: conditions — Infertility, Female | interventions — Growth Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GH group (Experimental): Growth Hormone adding to controlled ovarian hyperstimulation
  Interventions: Drug: Growth hormone
- control group (No Intervention): regular controlled ovarian hyperstimulation

INTERVENTIONS:
Drug: Growth hormone — GH has been considered as a cogonadotropin, which plays an important role in the synthesis of ovarian steroid hormone and follicular development as a paracrine hormone.GH can regulate the growth hormone receptor and strengthen the function of mitochondria to improve the quality of the female oocyte.
  Other Names: Experimental group
  Arms: GH group

SUMMARY:
GH plays an important role in the synthesis of ovarian steroid hormone and follicular development as a paracrine hormone.GH can regulate the growth hormone receptor and strengthen the function of mitochondria to improve the quality of the female oocyte.In this study, a prospective randomized control was used to explore the effect of GH adjuvant therapy on embryo quality.

ELIGIBILITY:
Inclusion Criteria:

* 1)infertility women whose age ≥20 and ≤39 years old; 2)women has done IVF/ICSI assisted treatment ≥1 times； 3)number of IVF/ICSI assisted treatment cylces with ≥6 oocytes retrieved ≥1； 4)number of IVF/ICSI assisted treatment cylces with ≥50% fertilization rate ≥1 ; 5)historical assisted reproduction cycles without ≥6C-Ⅱ level embryos at the third day after oocytes retrieval or without blastocyst formation after blastocyst culturing.

Exclusion Criteria:

- 1) Diseases related to IVF treatment outcome, such as untreated hydrosalpinx, uterine fibroids affecting uterine cavity, myometriosis, endometrial lesions, obvious uterine abnormalities,etc; 2)Severe acute or chronic liver or kidney diseases, such as cirrhosis, acute or chronic renal failure, hepatitis B virus activity period,etc.;in patients with abnormal liver and kidney function, the AST or ALT detection value was 2.5 times higher than the upper limit of normal, and the serum creatinine was 2 times higher than the upper limit of normal.

3)Endocrine and metabolic diseases and adrenal diseases, such as diabetes, Cushing's syndrome,etc.; 4)People has allergy history of growth hormone product; 5)Participating in other clinical research; 6)Other conditions that researchers determined not fit to be enrolled.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
number of high-quality embryos at D3 | the third day after oocyte retrieval
  number of embryos grading 6C-II and above 6C-II at the third day after oocyte retrieval
proportion of high-quality embryos at D3 | the third day after oocyte retrieval
  proportion of embryos grading 6C-II and above 6C-II at the third day after oocyte retrieval

SECONDARY OUTCOMES:
clinical pregnancy rate | 28 days after embryo transplanted
  proportion of patients with presence of a gestational sac with fetal heartbeat by transvaginal ultrasound at 28 days after ET in transplanted patients
number of high-quality oocytes | four months
  number of oocytes with diameter ≥18mm at triggering day
implantation rate | 28 days after embryo transplanted
  proportion of implanted embryos in transplanted embryos
total amount of Gn used | four months
  total amount of Gn used
total days of Gn used | two months
  total days of Gn used
E2 levels at triggering day | four months
  E2 levels at triggering day
IGF-I level at the first day of injecting GH and befor injecting GH(GH group) | at the first day of injecting GH and befor injecting GH(GH group)
  IGF-I level at the first day of injecting GH and befor injecting GH(GH group)
IGF-I level at the first day of injecting Gn and before injecting Gn | at the first day of injecting Gn and before injecting Gn
  IGF-I level at the first day of injecting Gn and before injecting Gn
IGF-I level at triggering day | four months
  IGF-I level at triggering day
number of blastocysts at the fifth,sixth or seventh day after oocyte retrieval | at the fifth,sixth or seventh day after oocyte retrieval
  number of blastocysts formation after culturing at the fifth,sixth or seventh day after oocyte retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Fei Gong, Doctor, Study Director — Reproductive & Genetic Hospital of CITIC-Xiangya
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China

REFERENCES:
- [Derived] Tang Y, Li X, Hu C, Guan R, Wang Z, Zhang S, Tao G, Qu J, Gong F. Exploring the potential benefits of growth hormone co-treatment on embryo quality in IVF: a randomized controlled open-label trial. Reprod Biol Endocrinol. 2025 Mar 15;23(1):42. doi: 10.1186/s12958-025-01374-3. PMID 40089744